CLINICAL TRIAL: NCT06468293
Title: The Role of Caregiver in the Clinical Pathway of Patients Newly Diagnosed With Breast and Prostate Cancer: a Randomized Study
Brief Title: Role of Caregiver in the Clinical Pathway of Patients With Breast and Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IEO 1702
Record Dates: First submitted 2024-03-26; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Non psychological support intervention
- Intervention group (Other): Psychological support intervention with scheduled appointment within the period of diagnostic assessment
  Interventions: Other: Psychological support

INTERVENTIONS:
Other: Psychological support — Psychological support intervention
  Arms: Intervention group

SUMMARY:
The following randomized longitudinal study will evaluate the long term impact of caregivers' involvement in cancer care pathway, including a psychological support intervention on the dyads to be delivered after the detection of a suspected cancer and before the visit with the oncologist for discussing therapeutic options.

DETAILED DESCRIPTION:
The following randomized longitudinal study will evaluate the long term impact of caregivers' involvement in cancer care pathway, including a psychological support intervention on the dyads to be delivered after the detection of a suspected cancer and before the visit with the oncologist for discussing therapeutic options. Moreover, a battery of self-report questionnaires will be administered, and sociodemographic and clinical data will be collected. The time window in which to deliver the support intervention is after the detection of a suspected cancer and before the visit with the oncologist, at the time when the patient undergoes diagnostic exams (to understand the type of tumor he/she is affected by), and the most suitable therapeutic protocol have to be discussed with the oncologist.

ELIGIBILITY:
Inclusion Criteria:

Patient:

* Patient aged ≥18 years at the time of recruitment.
* Patients who have just received a cancer diagnosis and have yet to discuss with their oncologist the treatment to undergo after diagnosis of breast or prostate cancer.
* Early-stage cancer (I or II).

Caregiver:

* Age ≥ 18 at the time of recruitment.
* Taking care of the patient.

Exclusion Criteria:

Patients:

* Presence of early mental disorders (before age 40) or severe neurological disorder.
* Patients with advanced stage cancer for which the path is already defined (palliative care patients).

Caregivers:

● Presence of early mental disorders (before age 40) or severe neurological disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2022-10-08 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the compliance with therapy | 6 months
  The primary endpoint of this study is to observe a difference of 3 points in the average values of the "Interpersonal aspect of care" and "Subjective norm" subscales of the Adherence Determination Questionnaire (ADQ), in favor of the intervention group.
  Response options for each item formed a 5-point Likert scale (1 = strongly disagree; 2 = disagree; 3 = neither agree nor disagree; 4 = agree; 5 = strongly agree). The ADQ questionnaire contains 38 questions, with items 15 and 17 through 24 specifically phrased for patients who have cancer

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Pravettoni, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy